CLINICAL TRIAL: NCT01461447
Title: Safety and Immunogenicity Following Further Boosting With HIV-1 MVA-CMDR Vaccine to HIVIS03 Volunteers Who Were Primed With HIV-1 DNA Low Dose Intradermally or 'Standard' Dose Intramuscularly and Boosted With MVA-CMDR Vaccine
Brief Title: Safety Study of an Additional MVA Vaccine in Volunteers Who Received 3 DNA Vaccines Followed by 2 MVA Vaccines
Acronym: HIVIS06
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Muhimbili University of Health and Allied Sciences (Other)
Collaborators: Karolinska Institutet (Other); Swedish Institute for Infectious Disease Control (Other); Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Patricia Jane Munseri, MD, Muhimbili University of Health and Allied Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: HIVIS 06
Record Dates: First submitted 2011-10-20; First posted 2011-10-28 (Estimated); Last update posted 2012-05-24 (Estimated); Status verified 2012-05

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — smallpox and monkeypox vaccine modified vaccinia ankara-bavarian nordic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MVA (Experimental): Volunteers who were primed with 3 HIVIS DNA and further boosted with 2 MVA vaccine will receive a third MVA there shall not be an comparator for this study.
  Interventions: Biological: Modified Vaccinia Ankara

INTERVENTIONS:
Biological: Modified Vaccinia Ankara — Healthy volunteers will receive intramuscularly 1 injection of MVA-CMDR 1ml (Total 10 power 8 pfu) boost injection in the left deltoid muscle.

SUMMARY:
The purpose of the study is to determine the safety and immunogenecity of a third MVA in the HIVIS 03 volunteers who have received 3 HIVIS DNA vaccines followed by boosting with 2 MVA vaccines.

The investigators postulate that the Immune responses that were observed in the HIVIS 03 trial are likely to wane over time. To date it is unknown how these responses should best be maintained. In this study the investigators seek to boost immune responses, especially the antibody responses induced by the second MVA boost.

Since the HIV specific antibodies were induced only after the second MVA injection, it is hypothesized that a 3rd MVA will give rise to even higher and sustained antibody titers.

ELIGIBILITY:
Inclusion Criteria:

1. Have completed the HIVIS03/TaMoVac01 WP1 protocol and received the active vaccine
2. Willing to undergo counseling and HIV testing
3. Are not infected by HIV infection as indicated by a negative PCR reaction against HIV.
4. Able to give informed consent
5. Resident in Dar es Salaam, and willing to remain so for the duration of the study
6. At low risk of HIV infection, defined as the absence of an identifiable risk factor/ behavior:

   * sexual partner with HIV
   * sexual partner with unknown HIV serostatus who is also unwilling to use protective condoms consistently in all sexual relations
   * sexual partner is known to be at high risk for HIV
   * more than one sexual partner in the last 6 months.
   * history of being an alcoholic [as medically defined or more than 35 units /week]
   * History of STI within past 6 months.
7. Verbal assurances that adequate birth control measures are used not to conceive/father a child during the study and up to 4 months after the 3rd MVA vaccine injection
8. Have a negative urinary pregnancy test for females
9. ECG findings that neither pose a risk for the vaccination nor preclude evaluation of peri/myocarditis.
10. Be willing to practice safe sex for the duration of the study to avoid sexually transmitted infections including HIV.
11. Good health as determined by medical history, physical examination, clinical judgment and by key laboratory parameters

Reference ranges will be in accordance with data generated at MUHAS for hematology values, and biochemical parameters. Exclusion by presence of Diabetes mellitus will be based on the WHO cut-off value of a Fasting Blood Glucose >7.8 mmol/l

No grade 1 or higher routine laboratory parameters (see section on appendix 3 DAIDS chart for Definitions). Hence lab parameters have to be as follows:

* Hb >10.5g/dl
* White blood cell count >1,300/mm3
* Lymphocytes >1.0/ mm3
* Platelets >120,000/ mm3
* CD4 >400cells/ mm3
* Random Blood Glucose 2.5-7.0 mmol/L; if elevated, then a Fasting Blood Glucose <7.8 mmol/l
* Bilirubin <1.25 x uln
* ALT <1.25 x uln
* Creatinine <1.25 x uln
* Urine dipstick for protein and blood: negative or trace. (If either is ≥ 1+, obtain complete urinalysis (UA). If microscopic UA confirms evidence of hematuria or if proteinuria ≥ 1+, the volunteer is ineligible).

Exclusion Criteria:

1. Active tuberculosis or other systemic infectious process elicited by review of systems, physical examination and laboratory detection. Such as detection of Hepatitis B surface antigen, or active syphilis.
2. Have a history of immunodeficiency, chronic illness requiring continuous or frequent medical intervention
3. Autoimmune disease by history and physical examination.
4. Severe eczema
5. Have history of psychiatric, medical and/or substance abuse problems during the past 6 months that the investigator believes would adversely affect the volunteer's ability to participate in the trial.
6. History of grand-mal epilepsy, or currently taking anti-epileptics
7. Have received blood or blood products or immunoglobulins in the past 3 months.
8. Are receiving immunosuppressive therapy such as systemic corticosteroids or cancer chemotherapy.
9. Have used experimental therapeutic agents within 30 days of study entry.
10. Have received any live, attenuated vaccine within 60 days of study entry. {NOTE: Medically indicated subunit or killed vaccines (e.g., Hepatitis A or Hepatitis B) are not exclusionary but should be given at least 2 weeks before or after HIV immunization to avoid potential confusion of adverse reactions}.
11. History of severe local or general reaction to vaccination defined as:

    * Local: Extensive, indurated redness and swelling involving most of the major circumference of the arm, not resolving within 72 hours
    * General: Fever >= 39.5 0C within 48 hours; anaphylaxis; bronchospasm; laryngeal oedema; collapse; convulsions or encephalopathy within 72 hours
12. Are lactating mothers
13. Are study site employees who are involved in the protocol and may have direct access to the immunogenicity results
14. Unlikely to comply with protocol as judged by the principal investigator or her designate.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-03; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Proportion of volunteers with humoral and cellular immune responses elicited by 2 different immunization schedules (id or im DNA priming) prior to MVA boosting | 1 month after vaccination
Safety assessed by the number of solicited and non solicited adverse events following immunization | 1 month after vaccination

SECONDARY OUTCOMES:
Number of staff trained and able to conduct HIV-related vaccine studies at MUHAS. | Two months

CONTACTS AND LOCATIONS:
Locations (1):
- Muhimbili University of Health and Allied Sciences, Dar es Salaam, Tanzania